CLINICAL TRIAL: NCT01172873
Title: Open-Label Exploratory Investigation of D-Cycloserine Augmentation to Cognitive Behavioral Therapy With Exposure and Response Prevention for Adults and Adolescents Diagnosed With Obsessive Compulsive Disorder - A Feasibility Study
Brief Title: D-Cycloserine Augmentation to CBT With Exposure and Response Prevention in Adults and Adolescents With OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #5828
Record Dates: First submitted 2009-04-20; First posted 2010-07-30 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; DCS; D-cycloserine; CBT; E/RP; exposure response prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCS + Exposure and Response Prevention (Active Comparator): Participants in this arm receive 10 twice-weekly 60-minute sessions of Exposure and Response Prevention (E/RP) therapy and 50mg of D-Cycloserine immediately after each therapy session. D-Cycloserine is only administered on days in which therapy sessions are held.
  Interventions: Drug: D-cycloserine; Behavioral: Exposure and Response Prevention (EX/RP)
- E/RP alone (no DCS administration) (Active Comparator): Participants in this arm received twice-weekly 60 minute sessions of E/RP alone for a total of 10 sessions.
  Interventions: Drug: D-cycloserine; Behavioral: Exposure and Response Prevention (EX/RP)

INTERVENTIONS:
Drug: D-cycloserine — 50 mg dose of D-cycloserine administered at the end of each session of Cognitive Behavioral Therapy With Exposure and Response Prevention: twice weekly CBT/ERP of 60 minutes
Behavioral: Exposure and Response Prevention (EX/RP) — Exposure and response prevention treatment. Participants complete graded exposure during twice weekly treatment sessions with therapist

SUMMARY:
This is a single site, open-label, feasibility study of cognitive behavioral therapy with exposure and response prevention (CBT/ERP) adding the augmentation of D-cycloserine (DCS) for adolescents ages 12-17 with Obsessive Compulsive Disorder (OCD) who are partial or non-responders to first line treatments of CBT or pharmacotherapy.

DETAILED DESCRIPTION:
The primary goal of this study is to examine the feasibility and efficacy of DCS augmentation to CBT/ERP at the end of the session. The main treatment outcome will be measured by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). The secondary goal of the study is to investigate the safety of DCS in adolescents with OCD. 18 adolescents will be recruited in this study. Patients who are currently on medication therapies for OCD must be stable for at least 12 weeks prior to and during the study.

This study consists of a screening period that contains a 90-minute psycho-educational session and treatment period of up to 5 weeks. During the treatment period, patients will receive ten 60-minute CBT/ERP sessions held twice weekly. At the end of each session, patients will receive a 50 mg dose of DCS. Following the administration of the DCS, patients will be asked to do their best not to ritualize and remain on the Children's Day Unit, where they will be observed and report to the research team if any ritualization has occurred. At the end of study participation, all participants will be offered 10 additional sessions of twice-weekly ERP without DCS administration. All participants will then complete a follow-up visit at 10 weeks after baseline.

The main treatment outcome will be measured by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). The secondary goal of the study is to investigate the safety of DCS in adolescents with OCD. Additionally, we will explore the impact of patient's motivation to change, parental pathology, and family accommodation on the treatment progress and outcome in adolescents.

Present data collected from this protocol show that adolescents who completed and engaged in treatment experienced benefit to the combination of CBT/ERP and DCS. However, this is an unblinded study and the adolescents are receiving an intensive form of CBT/ERP with close monitoring following 2 hours after the administration of the DCS. The positive results may be due to this specific way in which the CBT/ERP was delivered or to the attention paid to participants during treatment sessions and monitoring periods. We recruited 5 additional adolescents diagnosed with OCD to serve as control group participants. These individuals all had a history of failed or partial response to at least one trial of Selective Serotonin Reuptake Inhibitor (SSRI) medication or CBT/ERP. These participants also received ten sessions of twice weekly CBT/ERP delivered exactly as it was previously in this protocol, but without DCS administration. All control participants completed a follow-up visit at 10 weeks after baseline. Due to the small number of control participants, statistical analyses comparing the treatment groups were not completed.

ELIGIBILITY:
Inclusion/Exclusion Criteria

Inclusion Criteria:

1. Patients must be ages of 12-17 at the time of consent.
2. Both patients and parents must be able to speak and understand English.
3. Written informed assent by the patient and consent by the parent.
4. Ability and willingness to comply with study treatment and to attend study assessments.
5. Patients must be physically healthy males or non-pregnant females. Females of childbearing potential must comply with contraceptive restrictions noted in the protocol.
6. Patients must fulfill Diagnostic and Statistical Manual (DSM-IV) criteria for OCD, and OCD must be the primary disorder with a CY-BOCS score > 16
7. For patients with attention-deficit hyperactivity disorder (ADHD), the condition must be stable for 4 weeks on present treatment prior to screening.
8. For patients receiving treatment with an FDA approved Serotonin Reuptake Inhibitor (SRI), the medication dose must be stable for at least 12 weeks prior to enrollment.
9. Patients who failed to respond to either CBT/ERP treatment or a SRI medication (as evidenced by a CY-BOCS score > 16).
10. Based on history, the patient is unlikely to require a change in medication during the course of CBT/ERP + DCS treatment.

Exclusion Criteria:

1. Patients with any clinically significant abnormalities in laboratory parameters at screening.
2. Clinically significant metabolic-endocrine, hematological, gastrointestinal disease, pulmonary disease (for example, severe asthma, uncontrolled diabetes mellitus).
3. History of schizophrenia or any psychotic disorder, history of mental disorders or any present Axis I psychiatric disorder according to DSM-IV criteria (using the Anxiety Disorders Interview Schedule (ADIS-R) assessment interview), except for patients with a diagnosis of ADHD and/or other anxiety disorders as secondary diagnoses.
4. Patients who have a history suggestive of Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infection (PANDAS). - i.e., a sudden onset or exacerbation of symptoms temporally associated with a preceding streptococcal infection with first onset prior to puberty.
5. Patients who are receiving formal psychotherapy, other than the one delivered in the study, whether or not the focus of the therapy is on their OCD.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moira A Rynn, M.D., Principal Investigator — NYSPI / CU
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was drawn from the broadest possible population with respect to gender and ethnic origin. Internal Review Board(IRB)-approved web/radio/newspaper ads & flyers were used to recruit patients, as were physician and mental health practitioner referrals.
Pre-assignment Details: 16 adolescents(12-17yrs) participated in the study. The initial 11 participants received 10 twice-weekly sessions of exposure and response prevention treatment (E/RP) as well as D-Cycloserine(DCS) 50mg at each session. The final 5 participants received 10 twice-weekly sessions of E/RP treatment alone during the active study period.
Groups:
- D-cycloserine + E/RP: The first 11 participants received 10 twice-weekly 60-minute sessions of exposure and response prevention (E/RP) during the active study period. D-Cycloserine 50 mg was administered immediately after each therapy session.
- E/RP Alone (no DCS Administration): The final 5 participants enrolled in the study were assigned to a second treatment arm, to compare E/RP alone to E/RP with D-Cycloserine. These participants received 10 twice-weekly sessions of E/RP without D-Cycloserine. DCS was not administered to this group during the active study period.
Period: Overall Study
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration)
Started | 11 | 5
Completed | 8 | 3
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Sixteen participants ages 12-17 were enrolled in the study. All met criteria for a principal disorder of OCD. One participant consented but was then deemed ineligible to participate prior to baseline.
Groups:
- D-cycloserine + E/RP: Participants in this treatment arm received 10 twice-weekly sessions of E/RP treatment and were administered D-Cycloserine (DCS) immediately after every treatment visit.
- E/RP Alone (no DCS Administration): Five participants were enrolled in the second treatment arm as a comparison. The participants received 10 twice-weekly sessions of E/RP treatment alone.
- Total: Total of all reporting groups
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration) | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 5 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.67 (1.32) | 16.25 (.96) | 15.85 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS) for Adolescents
Description: The CYBOCS is a semi-structured measure of Obsessive Compulsive Disorder (OCD) severity with excellent inter-rater reliability, internal consistency, and test-retest reliability. It is validated in those starting at age 7 and used in studies up to age 20.The CYBOCS differs from the adult Yale-Brown Obsessive Compulsive Scale (YBOCS) only in its use of simpler language. CYBOCS scores range from 0-40, with higher scores representing greater severity of symptoms. The CYBOCS will be administered by independent evaluators (IEs) at baseline, session 5, session 10 and the follow-up visit. It will be the primary outcome measure. The CYBOCS checklist will be used to determine symptom dimensions.
Time Frame: baseline, visit 5, visit 10, follow-up visit
Population: Data from 14 adolescents were analyzed. One participant was excluded from analyses because he did not receive DCS at every treatment visit. Another was excluded because she was unable to provide reliable data on outcome measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- D-cycloserine + E/RP: Treatment involved 10 twice-weekly 60-minute sessions of exposure and response prevention (E/RP) during the active study period. D-Cycloserine 50 mg was administered immediately after each therapy session.
- E/RP Alone (no DCS Administration): Participants receiving 10 twice-weekly sessions of E/RP treatment alone. DCS was not administered to this group during the active study period.
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration)
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline CYBOCS | 26.56 (3.91) | 27.25 (3.6)
  Session 5 CYBOCS | 22.44 (5.17) | 19.8 (7.26)
  Session 10 CYBOCS | 19.67 (8.77) | 17.2 (11.55)
  Follow-Up CYBOCS | 14.5 (7.78) | 22 (3.61)

2. Secondary Outcome: Multidimensional Anxiety Scale for Children (MASC)
Description: Multidimensional Anxiety Scale for Children (MASC): This is a 39-item self-report that measures anxiety symptoms. It provides a total score, as well as 10 subscales, although only total scores will be analyzed. MASC scores range from 0-117, with higher scores representing greater severity of anxiety symptoms. The MASC and will be administered at baseline, session 5, session 10 and the follow-up visit for adolescents.
Time Frame: baseline, visit 5, visit 10, follow-up visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration)
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline MASC | 42.67 (23.37) | 52.4 (23.56)
  Session 5 MASC | 40.56 (19.79) | 47.4 (29.72)
  Session 10 MASC | 39.33 (21.42) | 46.8 (31.25)
  Follow-Up MASC | NA (NA) — Data were not collected at the follow-up visit for this treatment arm. | 40.5 (41.72)

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Beck's Depression Inventory (BDI): This is a 21-item self report that measures depression symptoms and will be used for both adults and adolescents at baseline, session 5, session 10 and the follow-up visit. BDI-II scores range from 0-63, with higher scores representing greater severity of depression symptoms.
Time Frame: baseline, visit 5, visit 10, follow-up visit
Population: Data from 14 adolescents were analyzed. One participant was excluded from analyses because he did not receive DCS at every treatment visit. Another was excluded because she was unable to provide reliable data on outcome measures. Another was excluded because she was unable to provide reliable data on outcome measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration)
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline BDI | 13.11 (12.41) | 12.5 (0.71)
  Session 5 BDI | 11.33 (8.23) | 4.8 (2.95)
  Session 10 BDI | 9.67 (7.21) | 4 (2.35)
  Follow-Up BDI | NA (NA) — Data were not collected at the follow-up visit for this treatment arm. | 4.34 (1.53)

ADVERSE EVENTS:
Groups:
- D-cycloserine + E/RP: Participants in this arm receive 10 twice-weekly 60-minute sessions of Exposure and Response Prevention (E/RP) therapy and 50mg of D-Cycloserine immediately after each therapy session. D-Cycloserine is only administered on days in which therapy sessions are held.
Arm/Group | D-cycloserine + E/RP | E/RP Alone (no DCS Administration)
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/5
Other Adverse Events (participants affected / at risk) | 6/11 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine + E/RP (N=11) | E/RP Alone (no DCS Administration) (N=5)
Worsening of OCD symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Worsening of OCD symptoms leading to inpatient hospitalization
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine + E/RP (N=11) | E/RP Alone (no DCS Administration) (N=5)
Headache (General disorders) | 3 (5) | 2 (3)
GI distress (Gastrointestinal disorders) | 2 (4) | 2 (2)
Exacerbation of anxiety (Psychiatric disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to small sample size of treatment groups, analyses comparing groups were not conducted. Therefore, we cannot conclude that findings were due to D-cycloserine (DCS) augmentation.

All participants received treatment from the same therapist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No